CLINICAL TRIAL: NCT02812732
Title: DOSE HPV: Development of Systems and Education to Improve HPV Vaccination Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Boston University (Other); American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Rebecca Perkins, Associate Professor, Boston Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: H-34561
Record Dates: First submitted 2016-06-21; First posted 2016-06-24 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Behavior
Keywords: HPV vaccination; provider education
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Providers at each clinic will receive the intervention (DOSE HPV) on a rolling basis. Vaccination rates will be compared pre- and post-intervention at each clinic, and changes in rates will be compared across clinics.
  Interventions: Behavioral: DOSE HPV

INTERVENTIONS:
Behavioral: DOSE HPV — The primary goals of the DOSE HPV intervention are to 1) change clinician HPV vaccine recommendations and responses to hesitant parents, and 2) support systems changes to improve the vaccination process. The first four sessions follow a standardized curriculum, while the last three sessions include development and implementation of tailored activities designed to meet individual practice needs.
  Sessions 1 and 2 generate motivation for the project through feedback of vaccination rates (Session 1) and education on HPV disease (Session 2). Brief Negotiated Interview (BNI) skills are taught in Sessions 3&4. Action Plans are developed in Session 5. Sessions 6&7, which follow a standard quality improvement format: plan-do-study-act (PDSA) cycles.

SUMMARY:
After completing over 600 interviews with parents, adolescents, and clinicians to determine reasons why HPV vaccines are used or not used, the investigators recently piloted a communication-based educational intervention with healthcare clinicians to improve communication around HPV vaccination. The intervention combined education and quality improvement methods using a mechanism called Performance Improvement Continuing Medical Education. This type of intervention is attractive to clinicians because they improve their cancer prevention practices while fulfilling requirements for maintaining board certification. The intervention consists of seven education and feedback sessions along with baseline and follow-up chart reviews and facilitated group discussions of clinician and practice vaccination rates. The pilot intervention was effective: at the two pilot intervention sites, girls were 60% and boys were 15 times more likely to receive HPV vaccination than at control sites both during and after the intervention period.

The goal of the proposed research is to broadly test the intervention's effectiveness in a diverse group of pediatric and family medicine practices serving low-income and minority patients. First, the investigators will perform a randomized trial in five community health centers to determine the effectiveness of the intervention. Second, the investigators will examine what made the intervention successful and identify barriers to sustainability with the goal of ensuring that the intervention can be successfully replicated in other settings. Third, the investigators will explore the effects of the intervention on parent-clinician communication by surveying parents and clinicians and observing clinical encounters when vaccination is discussed.

The proposed intervention represents an innovative and scalable model for promoting cancer prevention and screening activities by clinicians. Unlike programs that increase administrative burdens on busy clinicians, the proposed intervention allows clinicians to improve cancer prevention practices while simultaneously fulfilling requirements to maintain their board certification and improving the quality of cancer prevention care. It therefore has great potential for widespread dissemination.

DETAILED DESCRIPTION:
BACKGROUND

Human Papillomavirus (HPV) causes cervical, vaginal, vulvar, anal, and oral cancers, which disproportionately affect low-income and minority populations. Universal HPV vaccination has the potential to decrease burdens and to reduce disparities in these diseases. However, HPV vaccination rates for U.S. adolescents remain low. Clinician recommendation is the most important factor influencing HPV vaccine uptake; thus enhancing clinician communication about HPV vaccines is a critically important target for interventions to prevent cancer.

OBJECTIVE

In the past six years, the investigators' research has identified factors affecting HPV vaccine communication and utilization. the investigators recently piloted a communication intervention with clinicians, and at the two pilot intervention sites, girls were 60% and boys were 15 times more likely to receive HPV vaccination than at control sites both during and after the intervention period. The investigators aim to demonstrate the effectiveness of this intervention in a randomized trial, and to directly examine its effects on communication.

SPECIFIC AIMS

Aim 1. To evaluate intervention effectiveness on raising HPV vaccination rates using a stepped wedge randomized trial in federally qualified health centers.

Aim 2: To conduct a process evaluation that examines barriers and facilitators to intervention implementation and intervention sustainability, and to assess intervention fidelity.

Aim 3. To describe specific effects of the intervention on clinician-parent communication about HPV vaccination.

STUDY DESIGN

To address Aim 1, the investigators will perform a stepped wedge randomized trial in five community health centers to determine the effectiveness of the intervention. The intervention consists of a seven session Performance Improvement Continuing Medical Education (PI CME) program that employs HPV education and training in motivational interviewing to improve clinicians' HPV vaccine communication, and allows clinicians to improve the quality of vaccine care while fulfilling board certification requirements. To address Aim 2, the investigators will individually interview a selected group of providers and clinical leaders using the Promoting Action on Research Implementation in Health Services (PARiHS) model of process evaluation, and will analyze audio recordings of clinical interactions to measure intervention fidelity. Aim 3, an exploration of the intervention's effects on parent-clinician communication, will be conducted by surveying parents and clinicians and observing clinical encounters.

CANCER RELEVANCE

Rates of HPV related cancers have been increasing, but vaccination rates have remained stagnant since 2011. Recognizing the potential impact of HPV vaccination, the President's Cancer Panel stated in 2014 that raising HPV vaccination rates was a national priority. The proposed intervention represents an innovative and scalable model for promoting cancer prevention and screening activities by clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Receive primary care at intervention sites
* ages 9-26

Exclusion Criteria:

* do not receive primary care
* outside age range

Ages: 9 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 382 (Actual)
Dates: Start 2016-04; Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Intervention effectiveness on increasing HPV vaccination rates using a stepped wedge randomized trial in federally qualified health centers. | Outcomes are assessed up to 36 months from the start of the study.
  Compare pre- and post-intervention rates of HPV vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Perkins, MD, Principal Investigator — Boston Medical Center/ Boston University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Perkins RB, Zisblatt L, Legler A, Trucks E, Hanchate A, Gorin SS. Effectiveness of a provider-focused intervention to improve HPV vaccination rates in boys and girls. Vaccine. 2015 Feb 25;33(9):1223-9. doi: 10.1016/j.vaccine.2014.11.021. Epub 2014 Nov 24. PMID 25448095
- [Derived] Casey SM, Jansen E, Drainoni ML, Schuch TJ, Leschly KS, Perkins RB. Long-Term Multilevel Intervention Impact on Human Papillomavirus Vaccination Rates Spanning the COVID-19 Pandemic. J Low Genit Tract Dis. 2022 Jan 1;26(1):13-19. doi: 10.1097/LGT.0000000000000648. PMID 34928249
- [Derived] Perkins RB, Legler A, Jansen E, Bernstein J, Pierre-Joseph N, Eun TJ, Biancarelli DL, Schuch TJ, Leschly K, Fenton ATHR, Adams WG, Clark JA, Drainoni ML, Hanchate A. Improving HPV Vaccination Rates: A Stepped-Wedge Randomized Trial. Pediatrics. 2020 Jul;146(1):e20192737. doi: 10.1542/peds.2019-2737. Epub 2020 Jun 15. PMID 32540986
- [Derived] Perkins RB, Banigbe B, Fenton AT, O'Grady AK, Jansen EM, Bernstein JL, Joseph NP, Eun TJ, Biancarelli DL, Drainoni ML. Effect of a multi-component intervention on providers' HPV vaccine communication. Hum Vaccin Immunother. 2020 Nov 1;16(11):2736-2743. doi: 10.1080/21645515.2020.1747923. Epub 2020 May 13. PMID 32401592